CLINICAL TRIAL: NCT06381973
Title: Influence of Airway Clearance Techniques on Ventilation Distribution in the Lateral Posture in COPD and Healthy Individuals
Brief Title: Ventilation Distribution in COPD Patients During Breathing Exercises
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: William Poncin, PT, PhD (Other)
Responsible Party: Sponsor-Investigator, William Poncin, PT, PhD, Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Organization: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ELTGOL
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Healthy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ELTGOL_Physio (Active Comparator): ELTGOL + Manual pressure of the physiotherapist
  Interventions: Behavioral: ELTGOL_Physio
- ELTGOL_Auto (Active Comparator): ELTGOL performed autonomously
  Interventions: Behavioral: ELTGOL_Auto
- PEP (Active Comparator): Positive expiratory pressure (PEP)
  Interventions: Device: PEP
- 1L-Tidal-Breathing (Active Comparator): Tidal-breathing of 1 liter per breath
  Interventions: Behavioral: 1L-Tidal-Breathing
- Spontaneous Breathing (Active Comparator)
  Interventions: Behavioral: Spontaneous Breathing

INTERVENTIONS:
Behavioral: ELTGOL_Physio — The subject will be asked to slowly exhale with the glottis opened in the right lateral posture. The physiotherapist will accompany the subject by gently applying manual pressure on the chest wall and the abdomen during expiratory phases.
  Arms: ELTGOL_Physio
Behavioral: ELTGOL_Auto — The subject will be asked to slowly exhale with the glottis opened in the right lateral posture. The physiotherapist will not intervene in this arm.
  Arms: ELTGOL_Auto
Device: PEP — The subject will be asked to exhale through a positive expiratory pressure (PEP) device (Threshold PEP) while being in the right lateral posture.
  Arms: PEP
Behavioral: 1L-Tidal-Breathing — The subject will be asked to breath with a fixed tidal-breathing of 1 liter per breath (monitored via a spirometer) while being in the right lateral posture.
  Arms: 1L-Tidal-Breathing
Behavioral: Spontaneous Breathing — The subject will be asked to breath spontaneously while being in the right lateral posture.
  Arms: Spontaneous Breathing

SUMMARY:
ELTGOL (Slow Expiration with the Opened Glottis in the Lateral posture) is an airway clearance technique performed in the lateral decubitus position. This technique focuses on optimizing ventilation of the infralateral lung (when the subject is lying in the lateral posture) to enhance local air-liquid interaction. Previous studies on ventilation differences between the infra- and supralateral lungs were conducted on healthy, young, male subjects, without the application of thoracic or abdominal pressure.

This study aimed to assess ventilation distribution in right lateral recumbency in patients with chronic obstructive pulmonary disease (COPD), as well as healthy individuals, and investigate the impact of thoracic and abdominal manual pressures during ELTGOL on ventilation distribution.

DETAILED DESCRIPTION:
Electrical impedance tomography will be used to verify the effect of the lateral posture and associated breathing techniques in COPD and healthy individuals. The subjects will be placed in a standardised position before the measurements begin. The subjects will be placed in a right lateral recumbency position. The protocol comprises four manoeuvres, each interrupted by a short rest phase. Each subject will begin the experiment with the spontaneous ventilation manoeuvre in order to obtain the reference ventilation distribution. This will be followed by four other manoeuvres during which ventilation was measured: 1) using an spirometer to obtain a tidal volume of 1L, 2) performing the ELTGOL technique independently, 3) performing the ELTGOL technique assisted by manual pressures applied by a physiotherapist. 4) using a positive expiratory pressure (PEP) device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: No acute or chronic respiratory disease, normal lung function, non-smoker.
* Patients with COPD: forced expiratory volume at one second (FEV1) ≤ 80% predicted value, in stable state.

Exclusion Criteria:

* Healthy subjects: obesity (BMI > 35kg/m²); active or former smoker; severe scoliosis; cardiovascular or neuromuscular disease; active implant (cardiac pacemaker or an implantable cardioverter-defibrillator (ICD); thoracic skin lesion.
* Patients with COPD: obesity (BMI > 35kg/m²); severe scoliosis; severe cardiovascular disease; neuromuscular disease; active implant (cardiac pacemaker or an implantable cardioverter-defibrillator (ICD); thoracic skin lesion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Impedance variation using Electrical Impedance Tomography | 2 minutes during intervention
  Impedance change in the right and left lungs

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium